CLINICAL TRIAL: NCT04463667
Title: Impact of Exercise Intervention for Patients With Non-alcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Professor Chun-Jen Liu, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202002056RIND
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Fatty Liver; NAFLD
Keywords: NAFLED
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The investigators will collect all basic information including intrahepatic fat and fibrosis severity, and assign them to the exercise intervention group (n = 80) and the observation group (n = 20) after conditional screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The effects of exercise intervention on fatty liver (Experimental): The effects of exercise intervention on fatty liver and the improvement of the above-mentioned various metabolic indicators, including improvement of sleep patterns and changes of intestinal microflora.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Collect all basic information including intrahepatic fat and fibrosis severity, and assign them to the exercise intervention group (n = 80) and the observation group (n = 20) after conditional screening.

SUMMARY:
In Taiwan, with the westernization of eating habit and lifestyle, metabolic syndrome and non-alcoholic fatty liver (NAFLD) have become very important health issues. This project will therefore study the histological and clinical data of patients with non-alcoholic fatty liver disease and explore the impact of exercise intervention on the hepatic fatty infiltration of the patients. The research strategy will include (1) combining modern artificial big data collection technology to fully monitor the daily life, sleep and exercise patterns of the participants; (2) improving fatty liver and metabolic syndrome through trial-based exercise intervention; and (3) exploring the changes of sleep patterns and intestinal microflora in patients with metabolic liver disease after exercise intervention.

DETAILED DESCRIPTION:
Background & aims: In Taiwan, with the investigators sternization of eating habit and lifestyle, metabolic syndrome and non-alcoholic fatty liver (NAFLD) have become very important health issues. This project will therefore study the histological and clinical data of patients with non-alcoholic fatty liver disease and explore the impact of exercise intervention on the hepatic fatty infiltration of the patients. The research strategy will include (1) combining modern artificial big data collection technology to fully monitor the daily life, sleep and exercise patterns of the participants; (2) improving fatty liver and metabolic syndrome through trial-based exercise intervention; and (3) exploring the changes of sleep patterns and intestinal microflora in patients with metabolic liver disease after exercise intervention.

Materials & methods: The investigators will first retrospective collect clinical and histologic data of patients with biopsy proven NAFLD. Second, the investigators will establish a non-invasive fatty liver detection and staging platform at National Taiwan University Hospital. The investigators then plan to enroll 100 patients with non-alcoholic fatty liver from NTUH employees. The investigators will collect all basic information including intrahepatic fat and fibrosis severity, and assign them to the exercise intervention group (n = 80) and the observation group (n = 20) after conditional screening. After one year of exercise intervention, the investigators will analyze the effect of exercise on intrahepatic fat (main parameter: 20% reduction in intrahepatic fat; 30% achieved in the exercise intervention group; 5% achieved in the control group) and related metabolic syndrome indicators, and analyze different types of exercise Whether the intervention has different effects, and analyze the improvement of sleep pattern and intestinal microflora after exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* non-alcoholic fatty liver from NTUH employees

Exclusion Criteria:

* not suitable for exercise (severe cardiovascular disease or severe limb and joint disease), patients with inherited hyperlipidemia (diabetes> 300 mg / dL or low-density lipoprotein cholesterol> 190 mg / dL or cardiovascular disease has occurred before the age of 60 )event).
* women exclude pregnancy and breastfeeding.
* liver cancer, AFP> 20 ng/ml.
* alcohol and drug abusers.
* the use of steroids, sex hormones, immunosuppressants, radiation exposure and chemotherapy within 3 months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
20% reduction in intrahepatic fat | 24 weeks.
  We aim to evaluate whether active exercise can help reduce the fat content of the liver. After 24-week exercise intervention, the effect of exercise on the reduction of intrahepatic fat content in cases (active exercise) versus controls (no exercise) will be assessed by MRS/PDFF

SECONDARY OUTCOMES:
Improvement of intrahepatic fibrosis | 24 weeks
  We also aim to evaluate whether active exercise can help reduce the fibrosis of the liver. After 24-week exercise intervention, the effect of exercise on the reduction of intrahepatic fat content in cases (active exercise) versus controls (no exercise) will be assessed by Fibroscan examination.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Jen Liu, Doctor, Principal Investigator — Department of Internal Medicine, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu CH, Yen KC, Wang LY, Hsieh PL, Wu WK, Lee PL, Liu CJ. Automated Whole-Liver Fat Quantification with Magnetic Resonance Imaging-Derived Proton Density Fat Fraction Map: A Prospective Study in Taiwan. Gut Liver. 2025 Jul 15;19(4):617-626. doi: 10.5009/gnl240408. Epub 2025 Apr 1. PMID 40169393